CLINICAL TRIAL: NCT04268121
Title: Phase II Study to Evaluate the Efficacy of 12-month Neoadjuvant Chemotherapy in Terms of Disease-free Survival in Patients With Localized Digestive Neuroendocrine Carcinomas
Brief Title: Efficacy of Neoadjuvant Chemotherapy in Terms of DFS in Patients With Localized Digestive Neuroendocrine Carcinomas
Acronym: NEONEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Fondation ARCAD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEONEC D19-01
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Carcinoma; Digestive Cancer
Keywords: Neoadjuvant treatment; Adjuvant treatment
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Gastrointestinal Neoplasms | interventions — Neoadjuvant Therapy; Cisplatin; Etoposide; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase II and prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase II (Experimental): Prospective, open, multi center, one-arm, national phase II study evaluating the benefits in terms of disease-free survival (DFS) at 12 months after the administration of neoadjuvant treatment in patients with localized digestive neuroendocrine carcinomas
  Interventions: Drug: Neoadjuvant treatment
- Prospective cohort (Active Comparator): Evaluation of DFS at 12 months in patients who underwent surgery and received adjuvant chemotherapy
  Interventions: Drug: Adjuvant treatment

INTERVENTIONS:
Drug: Neoadjuvant treatment — 4 cycles of platinum-based chemotherapy (carboplatin or cisplatin) plus etoposide followed by surgery or chemoradiotherapy
  Other Names: cisplatin / cisplatinum; etoposide / vepesid; carbopatin / paraplatin
  Arms: Phase II
Drug: Adjuvant treatment — Surgery (before study entry) followed by 4 cycles of platinum-based chemotherapy (carboplatin or cisplatin) plus etoposide
  Other Names: cisplatin / cisplatinum; etoposide / vepesid; carbopatin / paraplatin
  Arms: Prospective cohort

SUMMARY:
NEONEC is a single-phase, phase II study evaluating the efficacy of the 12-month neoadjuvant chemotherapy in patients with locally differentiated digestive NEC. The recommended chemotherapy is based on the current reference combination of platinum (cisplatin or carboplatin) and etoposide (VP16). For anorectal locations, radiochemotherapy is proposed to avoid the morbidity of conventional surgery.

The objective of the study is to improve relapse-free survival (RFS) in NEC patients treated with neoadjuvant chemotherapy followed by surgery or chemoradiotherapy.

In parallel, we will perform a prospective cohort study with patients whose diagnosis is made during surgery, who have not received neoadjuvant treatment, and who are offered an adjuvant treatment of the same type (combination of platinum and platinum salts and etoposide).

DETAILED DESCRIPTION:
A total of 48 patients is to be included in phase II and 30 patients in prospective cohort during the inclusion period of phase II.

Phase II study treatment:

Neoadjuvant chemotherapy: Administration of 4 cycles of chemotherapy (3 months) with platinum based chemotherapy (carboplatin or cisplatin, at the choice of the investigator) + etoposide.

Surgery or chemoradiotherapy depending on the tumor localization (the irradiation modalities and associated chemotherapy treatment will be left to the discretion of the referring radiotherapists according to current recommendations for each localization).

Prospective cohort:

* Surgery (prior to study entry)
* Adjuvant chemotherapy : Administration of 4 cycles of chemotherapy (3 months) with platinum based chemotherapy (carboplatin or cisplatin, at the choice of the investigator) + etoposide.

ELIGIBILITY:
Inclusion Criteria:

Phase II

1. Histologically proven digestive CNE, (the WHO 2017 classification: poorly differentiated and Ki 67 > 20%),
2. Patients with localized CNE, without metastasis (computed tomography [CT], thoraco-abdominopelvic CT scan [TAP] according to RECIST 1.1; examinations performed no later than 21 days before starting the study treatment, possible locoregional lymph node involvement defined according to the TNM classification),
3. Positron emission tomography (PET) and CT for lymph node status and elimination of secondary visceral and/or bone disorders, 4. Resectable tumor, according to the consensus decision made during local multidisciplinary surgical consultation meeting,

5. Age ≥ 18 years, 6. Written informed consent obtained from the patient, willing and able to comply with the protocol, 7. Registration in a National Health Care System (Protection Universelle Maladie [PUMa] included), 8. For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study treatment.

Men and women are required to use a reliable and adequate birth control during the study (if applicable) during the period of treatment and during 6 months from the last treatment administration.

Prospective cohort

1. Patients with localized digestive CNE histologically proven on the operative specimen (the WHO 2017 classification: poorly differentiated and Ki 67> 20%),
2. Localized, without metastasis on computed tomography [CT], thoracoabdominopelvic CT scan [TAP] RECIST 1.1, and/or locoregional lymph node involvement,
3. Age ≥ 18 years,
4. Written informed consent obtained from the patient, willing and able to comply with the protocol,
5. Registration in a National Health Care System (PUMa - Protection Universelle Maladie included),
6. For female patients of childbearing potential, negative pregnancy test within 7 days before starting the study treatment.

Men and women are required to use a reliable and adequate birth control methods during the study (if applicable) during the period of treatment and during 6 months from the last treatment administration.

Exclusion Criteria:

Phase II

1. Well-differentiated NEC, whatever the grade,
2. Metastatic disease,
3. Cancer of unknown primary
4. Organ failure that does not allow chemotherapy treatment,
5. Previous malignancy within 5 years prior to the study except for cutaneous basal cell carcinoma and uterine cancer in situ
6. Tumor with a mixed component (component accounts for ≥ 30%),
7. Patient impossible to follow-up,
8. Other than platinum-etoposide chemotherapy administrated,
9. Tutelage or guardianship or patient protected by law

Prospective cohort

1. Well-differentiated NEC, whatever the grade,
2. Metastatic disease,
3. Cancer of unknown primary
4. Organ failure that does not allow chemotherapy treatment,
5. Previous malignancy within 5 years prior to the study except for cutaneous basal cell carcinoma and uterine cancer in situ
6. Tumor with a mixed component (component accounts for ≥ 30%),
7. Patient impossible to follow-up,
8. Other than platinum-etoposide chemotherapy administrated,
9. Tutelage or guardianship or patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) - phase II | At 12 months
  Interval between the date of the start of treatment (chemotherapy) and the date of first relapse or death (all causes). Relapse is defined according to RECIST version 1.1 criteria.
Relapse-free survival (RFS) - prospective cohort | At 12 months
  Interval between the date of the start of treatment (chemotherapy) and the date of first relapse or death (all causes). Relapse is defined according to RECIST version 1.1 criteria.

SECONDARY OUTCOMES:
Number of patient in response in pre-operative or prior radiochemotherapy (if applicable) - Phase II | At 3 months after the beginning of treatment (up to 36 months)
  according to RECIST 1.1
Number of patients who do not benefit from surgery or radiochemotherapy (if applicable) - Phase II | Up to 39 months
  Number of patients who do not benefit from surgery or radiochemotherapy (if applicable) - Phase II
Number of patients operated after neoadjuvant chemotherapy or receiving radiochemotherapy (if applicable) - Phase II | Up to 39 months
  Number of patients operated after neoadjuvant chemotherapy or receiving
Overall survival (OS) - Phase II | up to 48 months
  Overall survival (OS) is defined as the time from study enrollment to death (from any cause) or to the last date the patients was known to be alive.
Overall survival (OS) - Prospective cohort | Up to 48 months
  Overall survival (OS) is defined as the time from study enrollment to death (from any cause) or to the last date the patients was known to be alive.
Number of participants with treatment-related adverse events grade 3-4 as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0 - Phase II | Up to 43 months
  Patients will be assessed for AEs throughout the study at every visit during treatment. Investigators using the NCI-CTCAE version 5.0 will grade the severity of AEs.
  Institute Common Terminology Criteria for Adverse Toxicity Study (NCI-CTCAE) version 5.0
Number of participants with treatment-related adverse events grade 3-4 as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0 - Prospective cohort | Up to 43 months
  Patients will be assessed for AEs throughout the study at every visit during treatment. Investigators using the NCI-CTCAE version 5.0 will grade the severity of AEs.
  Institute Common Terminology Criteria for Adverse Toxicity Study (NCI-CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Anna PELLAT, Principal Investigator — Saint-Antoine Hospital
Locations (14):
- France (14):
  - CHU Amiens - Hôpital Sud, Amiens
  - CHU Jean Minjoz, Besançon
  - Hôpital Beaujon, Clichy
  - CHU Dijon, Dijon
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Saint Antoine Hospital, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Haut Lévêque CHU Bordeaux, Pessac
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No